CLINICAL TRIAL: NCT04912479
Title: Can Connected Devices Increase the Success Rate of Benzodiazepine Withdrawals in the Elderly?
Acronym: BENZO-E-STOP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/19/0508; 2020-A02654-35 (Other: ID RCB)
Record Dates: First submitted 2021-05-28; First posted 2021-06-03 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Benzodiazepine Withdrawal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (No Intervention): Patients will be given a plan to reduce progressively their dosage of Benzodiazepin every 2 weeks. Over a 6-month period they will receive a phone call from the hospital twice a month to reinforce their motivation.
- intervention group (Experimental): In addition to the progressive withdrawal of BZD, patients will be given a connected watch that provide them with information on their sleep quality and their performed activities. They will also receive a check-up phone call twice a month over a 6-month period.
  Interventions: Device: connected watch

INTERVENTIONS:
Device: connected watch — connected watch that provide to patients with information on their sleep quality and their performed activities
  Arms: intervention group

SUMMARY:
This is a prospective randomized open study, which aims to evaluate the benefit of a connected watch to help people aged 65 years and older to withdraw from BZD over a six-month period, compared with classical withdrawal (e.g without connected watch). The study will include 100 patients, 50 in the control group and 50 in the intervention group.

Participants will be identified during a 12-month period through either external geriatric consultations or during a brief hospitalisation.

DETAILED DESCRIPTION:
Despite a trivialized use of benzodiazepine (BZD) in elderly people (EP), long-term efficacy is often questioned, and treatment has to be regularly re-examined to avoid side effects. Typical intervention techniques to aid patients in reducing their dosage involve: providing information about BZD, explaining the risks associated with a chronic exposure, and tips for a successful withdrawal. In addition, the usage of a connected device may reinforce the patient's motivation by providing details on the quality of sleep and the number of steps taken (activity).

This is a prospective randomized open study, which aims to evaluate the benefit of a connected watch to help people aged 65 years and older to withdraw from BZD over a six-month period, compared with classical withdrawal (e.g without connected watch). The study will include 100 patients, 50 in the control group and 50 in the intervention group.

Participants will be identified during a 12-month period through either external geriatric consultations or during a brief hospitalisation.

ELIGIBILITY:
Inclusion Criteria:

* Unassisted mobility (1/1 for the locomotion item on KATZ Activities of Daily Living scale)
* Mini-Mental State Examination (MMSE) ≥ 20
* With a daily consumption of benzodiazepine for more than 3 months
* Smartphone and/or tablet with internet connection

Exclusion Criteria:

* Patient under legal protection
* Patient refuses to participate
* Patient does not speak French

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-10-14 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
success to stop or reduce benzodiazepine consumption | 6 months
  success to stop benzodiazepine consumption (no more intake) or reduce benzodiazepine consumption (decrease in dosage of more than 25% or non-daily intake)

CONTACTS AND LOCATIONS:
Overall Officials: Cécile McCambridge, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No